CLINICAL TRIAL: NCT03990038
Title: Comparison of Two Multimodal Analgesia Regimens for Total Knee Arthroplasty : a Randomized Controlled Trial
Brief Title: Comparison of Two Multimodal Analgesia Regimens in Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems making the study completion unlikely
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, Principal investigator, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MultimodalTKA
Record Dates: First submitted 2019-06-15; First posted 2019-06-18 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone

STUDY DESIGN:
Intervention Model Description: Two multimodal analgesic protocols will be compared. Patients will be randomized to one of two analgesic protocol:
  C: Single-shot adductor canal block followed by a 48h perineurial continuous infusion of ropivacaine U: Single-shot adductor canal block and post operative extended release hydromorphone for 48h (4 doses)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants won't know their group because this study will use a double placebo:
  Group U: placebo for extended release hydromorphone (4 doses) Group C: sham perineurial infusion for 48h in group C (Perineurial catheter is connected to perineurial infusion pump but not infusion) Perineural infusion pumps will be covered with an opaque plastic bag to ensure blinding for patients and care providers Nurses and anesthesiologist and physiotherapist will be blinded to patient group allocation Investigator and outcome assessor will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group C (Active Comparator): Adductor canal block performed in the pre-operative period with 20 mL of Ropivacaïne 0.5%, followed with a continuous perineural infusion of Ropivacaïne 0.2%, 5 ml/h for 48 hours via a perineural catheter.
  They will also receive a placebo of Hydromorph Contin 3 mg, administered twice daily for 48h, starting on the evening after surgery
  Interventions: Drug: Continuous perineural infusion of ropivacaine 0.2% 5 ml/h for 48 h
- Group U (Active Comparator): Adductor canal block performed in the pre-operative period with 30 mL of Ropivacaïne 0.5%. A catheter is inserted in the adductor canal but no perineurial infusion. The catheter is connected to a pump that is shut down.
  They will also receive Hydromorph Contin 3 mg PO administered twice daily for 48 h, starting on the evening after surgery. 4 doses total
  Interventions: Drug: Extended Release Capsule

INTERVENTIONS:
Drug: Continuous perineural infusion of ropivacaine 0.2% 5 ml/h for 48 h — Group C receive the intervention Group U receives the placebo See arm description
  Other Names: Continous naropin infusion
  Arms: Group C
Drug: Extended Release Capsule — Group C receives a placebo for extended release hydromorphone Group U receives Hydromorph Contin 3 mg PO BID
  See arm description
  Other Names: Hydromorph Contin 3 mg PO BID for 48 h
  Arms: Group U

SUMMARY:
The improvement of postoperative analgesia is an important issue in orthopedic surgery, especially after total knee arthroplasty The use of a peripheral nerve block such as the adductor canal block is favored since it offers a postoperative analgesia superior to opioids, and also preserves the strength of the quadriceps, as opposed to the femoral block.

The adductor canal block can be given as a single injection (single shot) or a continuous perineural infusion to extend the block's analgesic duration. It is unclear if the continuous infusion is superior to the single shot. Indeed, a high catheter dislodgement rate is observed for this location and local anesthetics could migrate into the femoral canal, resulting in quadriceps weakness. Alternatively, adequate postoperative analgesia has been shown effective with a single shot adductor canal block combined with extended release opioids.

The primary objective in this study is to compare two analgesic protocols on the pain score at walk 24 hours after total knee arthroplasty.

Here are the two protocols compared :

1. Adductor canal block followed by continuous perineural perfusion for 48 hours
2. Adductor canal block (single shot) followed by hydromorphone extended release formulation for 48 hours In addition to analgesic adjuvants administered in both groups : acetaminophen, celecoxib, pregabalin, dexamethasone and periarticular infiltration.

Our hypothesis is that both protocols ensure a similar analgesia.

DETAILED DESCRIPTION:
The improvement of postoperative analgesia is an important issue in orthopedic surgery, especially after total knee arthroplasty. The early postoperative mobilization of these patients is crucial to ensure a favorable functional evolution, and this goal can't be accomplished without effective analgesia. Opioids offer an efficient pain relief, but their consumption can result in side effects that can increase the length of hospital stay. The use of a peripheral nerve block, such as the adductor canal block (BCA) is a widely favored alternative since it allows postoperative analgesia superior to opioids while preserving the strength of the quadriceps.

For a long period of time, the femoral block has been the most popular peripheral nerve block for patients after a knee arthroplasty. However, this perineural block is associated with an important rate of quadriceps' weakness, which could impair the post-operative mobilization and expose the patient to a risk of falling. It has now been widely replaced by the adductor canal block. The latter has the advantage of providing analgesia at rest and during movement equivalent to the femoral block, while preserving the quadriceps strength and offering a better mobility in the first 24 hours after surgery. In opposition to the femoral block, the adductor canal block does not increase the risk of falling since it is mainly a sensitive block.

The adductor canal block is an advantageous analgesic modality for patients after TKA, but it is limited since it offers only analgesia to the anteromedial aspect of the knee, sparing the lateral and posterior faces. It is common to combine this block with a periarticular knee infiltration with local anesthetics, performed by the surgical team at the end of the surgery. The two modalities combined make it possible to achieve very low pains scores at rest and during walking, compared to both techniques used separately.

The adductor canal block can be administered in one unique injection or with a perineural continuous infusion, to extend the block's analgesic duration. However, it is uncertain whether there is an advantage to use a continuous infusion. There is a significant rate of catheter migrating out of the adductor canal and losing effect. There is also the possibility that the continuous infusion results in a proximal extent of local anesthetic in the femoral canal, generating quadriceps weakness that invalidates the benefits for ACB in the context of postoperative mobilization.

Indeed, the location of the catheter near the surgical site predisposes it to be dislodged out of the adductor canal during surgical manipulations in a significant proportion of patients. A rate as high as 30% of catheter dislodgement on postoperative day 1 was observed. It is possible to perform the block after surgery, before the dressing is applied, but this practice tends to create delays, which are not desirable in the actual context of optimization of the OR time.

In addition, perineural catheters require a strict surveillance by a specialized team and could interfere with patient mobilization because of the restriction associated with the equipment involved. It is reasonable to think that the absence of a catheter and an infusion pump offers an easier mobilization, although this has not been validated in clinical trials.

Finally, continuous infusions increase the cumulative dose of local anesthetics that the patients is exposed to. In order to reduce the toxicity risk, it is necessary to reduce the periarticular infiltration doses, which could impair the quality of analgesia.

Alternatively, it has been demonstrated that adequate post-operative analgesia could be obtained with an adductor canal block, combined with extended release opioids. Several clinical trials involving patients after total knee arthroplasty have shown that there is a benefit to using extended release opioids added to a multimodal analgesia protocol. Their pharmacokinetic profile ensures a more constant analgesia, while offering a safety profile similar to immediate release opioids, a lesser risk of respiratory depression and overdose. The usage of extended release opioids after TKA is justified since patients accuse moderate to severe pain during the first days after surgery, despite the use of a multimodal analgesia protocol and sustained consumption of immediate release opioids.

These two protocols have not been compared.

In conclusion, there is a consensus that postoperative analgesia in patients after TKA should be addressed with a multimodal analgesia protocol that includes a perineural block and analgesic adjuvants. However, the optimal composition of this protocol is not well defined. In our hospital center, the postoperative analgesia protocol for TKA includes a continuous adductor canal block for 48 hours, intravenous dexamethasone, periarticular infiltration of the posterior capsule by the surgeon and analgesic adjuvants such as acetaminophen, celecoxib and pregabalin.

Study outcome and hypothesis

The primary objective in this study is to compare two analgesic protocols on the pain score while walking 24 hours after total knee arthroplasty.

Here are the two protocols compared :

1. Adductor canal block followed by continuous perineural perfusion for 48 hours
2. Adductor canal block (single shot) followed by hydromorphone extended release formulation for 48 hours In addition to analgesic adjuvants administered in both groups : acetaminophen, celecoxib, pregabalin, dexamethasone and periarticular infiltration.

Our hypothesis is that both protocols ensure a similar analgesia.

Our secondary issues are the proportion of patient that achieve a pain score at walk < 4, the time for the 10 m walk test, the incidence of drowsiness, nausea and vomiting and the postoperative opioid use at 24 and 48 hours postoperatively.

This clinical trial is relevant since it aims to answer a frequently asked question in clinical practice, and its outcome will have a direct impact on the anesthetic practice. In addition, it aims to improve early postoperative mobilization with acceptable pain, which is important after orthopedic surgery.

Methodology

Study design This will be a prospective, randomized, double blind study.

Population Patients undergoing elective TKA

Duration of study 18 months

Sample size Assuming a walking pain score at day 1 of 4.8 (± 2.3) with continuous infusion adductor canal block, periarticular infiltration and analgesic adjuvants, 69 patients per group will detect a difference of 25% between pain scores in both groups, with a power of 90% and an alpha = 0.05. In order to compensate for the losses at follow-up, a total of 150 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old
* American Society of Anesthesiology physical status I-III
* Primary total knee arthroplasty surgery under regional anesthesia

Exclusion Criteria:

* Chronic kidney disease (CKD) with eGFR < 60mL/min
* Contraindications for the use of spinal anesthesia or adductor canal block : infection, sepsis, evolutive neurological disease, coagulopathy, patient refusal.
* Chronic use of opioids (>30 mg daily morphine equivalent)
* Documented allergy to Hydromorphone, tramadol, celecoxib, ropivacaine, pregabalin, acetaminophen and/or ketorolac
* Patient weight < 50 kg or BMI > 40
* Severe cardiac disease
* Severe pulmonary disease
* Chronic use of monoamine oxydase inhibitors
* Pregnancy
* Inability to give informed consent
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Pain score during walking (24 hours) | 24 hours postoperatively
  Verbal Numeric Scale pain score (0-10, where 0= no pain and 10= worst conceivable pain) during walking

SECONDARY OUTCOMES:
Pain score during walking (48 hours) | 48 hours postoperatively
  Verbal Numeric Scale pain score (0-10, where 0= no pain and 10= worst conceivable pain) during walking
Pain score at rest (24 hours) | 24 hours postoperatively
  Verbal Numeric Scale pain score (0-10, where 0= no pain and 10= worst conceivable pain) at rest
Pain score at rest (48 hours) | 48 hours postoperatively
  Verbal Numeric Scale pain score (0-10, where 0= no pain and 10= worst conceivable pain) at rest
Pain score at knee flexion (24 hours) | 24 hours postoperatively
  Pain score (Verbal Numeric Scale (0-10, where 0= no pain and 10= worst conceivable pain) at knee flexion
Pain score at knee flexion (48 hours) | 48 hours postoperatively
  Pain score (Verbal Numeric Scale (0-10, where 0= no pain and 10= worst conceivable pain) at knee flexion
Degree of knee flexion (24 hours) | 24 hours postoperatively
  Knee flexion (degrees) measured using a goniometer. More degrees indicates better knee flexion
Degree of knee flexion (48 hours) | 48 hours postoperatively
  Knee flexion (degrees) measured using a goniometer. More degrees indicates better knee flexion
10 minutes walking test (24 hours) | 24 hours postoperatively
  Number of meters walked during a 10 minutes period.
10 minutes walking test (48 hours) | 48 hours postoperatively
  Number of meters walked during a 10 minutes period
Incidence of Postoperative Nausea (24 hours) | 24 hours postoperatively
  number of patients experiencing postoperative nausea
Incidence of Postoperative Vomiting (24 hours) | 24 hours postoperatively
  number of patients experiencing postoperative vomiting
Incidence of Postoperative Nausea (48 hours) | 48 hours postoperatively
  Number of patients experiencing postoperative nausea
Incidence of Postoperative Vomiting (48 hours) | 48 hours postoperatively
  Number of patients experiencing postoperative vomiting
sedation score(24 hours) | 24 hours postoperatively
  Degree of sedation experienced by patients using a sedation scale score (0-3, where 0 = awake, no sedation, 3= asleep, impossible to arouse).
sedation (48 hours) | 48 hours postoperatively
  Degree of sedation experienced by patients using a sedation scale score (0-3, where 0 = awake, no sedation, 3= asleep, impossible to arouse).)
QoR-40 (48 hours) | 48 hours postoperatively
  Measurement of quality of recovery using the QoR-40 questionnaire. A greater score indicates better recovery profile
Cumulative opioïd dose (24 hours) | 24 hours postoperatively
  Cumulative dose of hydromorphone (milligrams) consumed for postoperative pain
Cumulative opioïd dose (48 hours) | 48 hours postoperatively
  Cumulative dose of hydromorphone (milligrams) consumed for postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Brulotte, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Ciusss, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No